CLINICAL TRIAL: NCT00197912
Title: Vaccination With Autologous Dendritic Cells Pulsed With Tumor Antigens for Treatment of Patients With Malignant Melanoma. Phase I/II Study
Brief Title: Dendritic Cell Based Therapy of Malignant Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Inge Marie Svane, MD, PhD, Department of Oncology, Herlev Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM0413
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2009-07

CONDITIONS: Advanced Melanoma
Keywords: dendritic cell; cancer vaccine; cyclophosphamide; melanoma
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide; Celecoxib; Interleukin-2; aldesleukin

INTERVENTIONS:
Biological: tumor antigen loaded autologous dendritic cells — DC vaccination regime consists of primary 10 intradermal injections of 1-2 weeks interval (q1w x 4 → q2w x 6). HLA-A2 positive patients are treated with p53, survivin and telomerase peptide-pulsed dendritic cells, and HLA-A2 negative patients are treated with allogeneic tumor lysate pulsed dendritic cells. 50 mg cyclophosphamide (Sendoxan®, Baxter A/S) is administered p.o. twice a day bi-weekly and 200 mg celecoxib (Celebra®, Pfizer) is given p.o. every day. From the 2nd vaccine, 2 MIU Interleukin-2 is administered s.c. on day 2-6.
  Other Names: Dendritic cell vaccine; Cyclophosphamide, Sendoxan®, Baxter A/S; Celecoxib, Celebra®, Pfizer; Interleukin-2, Proleukin®, Chiron B.V.

SUMMARY:
The aim of the study is to show if vaccination with autologous dendritic cells pulsed with peptides or tumor lysate in combination with adjuvant cytokines and Cyclophosphamide can induce a measurable immune response in patients with metastatic malignant melanoma, and to evaluate the clinical effect (objective response rate) of the vaccination regime.

DETAILED DESCRIPTION:
Eligible patients receive vaccination with tumor antigen pulsed autologous monocyte-derived mature dendritic cells with a fixed interval. The dendritic cells are generated from leukapheresis products and frozen after antigen loading.

HLA A2 positive patients are treated with PADRE and oncopeptide pulsed DC; p53, survivin and telomerase peptides. HLA A2 negative patients are treated with KLH and tumorlysate pulsed DC; autologous or allogeneic. Each patient is given 6 immunizations with at least 5x106 peptide/lysate pulsed autologous DC. Vaccination 1-4 is given weekly and 4-6 at 2-week intervals. Those patients who exhibit stable disease, partial response or complete response after 6 injections will be given 4 more vaccinations at 2-week interval. The vaccine is applied by intradermal injection near the inguinal region.

IL-2 2 MIU s.c. day 2-6, Cyclophosphamide (Sendoxan®, Baxter A/S) 50 mg twice a day bi-weekly and 200 mg Celecoxib (Celebra®, Pfizer) daily are used. Scans and re-staging tests are performed at scheduled intervals throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven progressive metastatic or locally advanced melanoma
* No standard treatment indicated
* Age: > 18
* WHO-Performance Status 0-1
* At least tone measurable tumor lesions according to the RECIST criteria.
* Life expectancy more than 3 months
* Acceptable CBC and blood chemistry results
* Written informed consent

Exclusion Criteria:

* Patients with a history of any other neoplastic disease less than 5 years ago (excepting treated carcinomas in situ of the cervix and basal/squamous cell carcinomas of the skin).
* Patients with metastatic disease in the central nervous system (CNS).
* Patients with other significant illness including severe allergy, asthma, angina pectoris or congestive heart failure.
* Patients with acute or chronic infection including HIV, hepatitis and tuberculosis.
* Patients who are pregnant.
* Patients who have received antineoplastic therapy including chemotherapy or immunotherapy less than 4 weeks before beginning the trial.
* Patients who receive corticosteroids or other immunosuppressive agents.
* Baseline serum LDH greater than 2.5 times the upper limit of normal.
* Patients with active autoimmune diseases such as lupus erythematosus, rheumatoid arthritis or thyroiditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Primary aim of the study is to evaluate tolerability and safety of the treatment | weekly the first four weeks thereafter biweekly

SECONDARY OUTCOMES:
Secondary aims: evaluation of treatment induced immune response and clinical response. | after 8 and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, MD, PHD, Principal Investigator — Department of Oncology, Copenhagen University Hospital, Herlev, Herlev Ringvej 75, DK-2760 Herlev, Denmark
Locations (1):
- Department of Oncology, Copenhagen University Hospital, Herlev, Herlev, Denmark

REFERENCES:
- [Background] Svane IM, Pedersen AE, Johnsen HE, Nielsen D, Kamby C, Gaarsdal E, Nikolajsen K, Buus S, Claesson MH. Vaccination with p53-peptide-pulsed dendritic cells, of patients with advanced breast cancer: report from a phase I study. Cancer Immunol Immunother. 2004 Jul;53(7):633-41. doi: 10.1007/s00262-003-0493-5. Epub 2004 Feb 25. PMID 14985857
- [Derived] Ellebaek E, Engell-Noerregaard L, Iversen TZ, Froesig TM, Munir S, Hadrup SR, Andersen MH, Svane IM. Metastatic melanoma patients treated with dendritic cell vaccination, Interleukin-2 and metronomic cyclophosphamide: results from a phase II trial. Cancer Immunol Immunother. 2012 Oct;61(10):1791-804. doi: 10.1007/s00262-012-1242-4. Epub 2012 Mar 20. PMID 22426890